CLINICAL TRIAL: NCT04226495
Title: Sufentanil Infusion vs Sufentanil Bolus and Time to Extubation During Routine Cardiac Surgery
Brief Title: Sufentanil Infusion vs Sufentanil Bolus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0520-20-FB
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sufentanil Bolus (Active Comparator): medication in scheduled doses (bolus)
  Interventions: Drug: Sufentanil Bolus
- Sufentanil Infusion (Experimental): medication in a slow trickle (infusion)
  Interventions: Drug: Sufentanil Infusion

INTERVENTIONS:
Drug: Sufentanil Infusion — Intra-operative sufentanil infusion
  Other Names: Sufentanil
  Arms: Sufentanil Infusion
Drug: Sufentanil Bolus — Intra-operative sufentanil bolus
  Other Names: Sufentanil
  Arms: Sufentanil Bolus

SUMMARY:
Randomized single blind controlled clinical trial to test the benefit of sufentanil infusion over bolus dosing to reduce time to extubation and reduced length of ICU stay.

DETAILED DESCRIPTION:
This study will compare Sufentanil bolus vs infusion and analyze which has a faster extubation time in participants who undergo routine cardiac surgery. The hypothesis is that routine cardiac surgery patients receiving sufentanil infusion will have a lower sufentanil concentration at the end of surgery and have a shorter time to extubation than participants receiving sufentanil bolus dosing even with similar total doses of sufentanil. The intervention will be Sufentanil infusion during surgery and evaluations will include Sufentanil blood concentrations, ICU and hospital length of stay and re-intubation rate. We will follow up with the participants through their ICU stay (primary objective) and hospital length of stay (secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled non-emergency cardiac surgical patients including those with planned procedures of CABG, AVR, and combined CABG and AVR
* 19 to 80 years old
* Planned pre-operative anesthesia screening visit and/or preoperative surgical clinic visit.
* Inpatient subject that is scheduled (greater than 24hrs in advance) for a non-emergency cardiac surgical case

Exclusion Criteria:

* Sufentanil allergy
* EF less than or equal to 30%
* Moderate or severe right ventricular dysfunction,
* Moderate pulmonary dysfunction, to include patients with at home 02 and/or daily bronchodilator therapy.
* End Stage Renal Disease on Dialysis
* Chronic Kidney Disease with GFR <30
* Sternotomy Re-do
* Emergency surgery
* Greater than 4 units of RBCs or FFP combined
* Mechanical circulatory support post-operatively such as ECMO, IABP, Impella
* Not eligible for rapid wean extubation protocol
* Requires infusion of sedative medication required during ICU admission
* Greater than or equal to 15 minute ICU hold within PACU

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Songster, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil Bolus | Sufentanil Infusion
Started | 32 | 33
Completed | 26 | 26
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 3 | 3
Not completed — PI discretion | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil Bolus | Sufentanil Infusion | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.4) | 63.3 (8.9) | 64.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Time to Extubation
Description: We will determine if sufentanil infusion administration intra-operatively during routine cardiac surgery will decrease time to extubation from OR stop data collection time point by 60 minutes compared to sufentanil bolus administration.
Time Frame: Amount of time in minutes from procedure finish to time of extubation, up to 800 minutes.
Population: The participant number represent the number of participant whom made it to this portion of the study.
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Sufentanil Bolus | Sufentanil Infusion
Number analyzed (Participants) | 26 | 26
Minutes | 230.5 [52 to 794] | 242.4 [58 to 691]

2. Secondary Outcome: Plasma Concentration
Description: We will determine if sufentanil infusion administration intra-operatively during routine cardiac surgery will result in a lower plasma concentration of sufentanil at time of arrival to ICU and if the plasma concentration correlates with time to extubation.
Time Frame: Lab concentration is drawn when patient arrives to ICU, an average of 1 hour after procedure.
Population: Lab concentration was measured on arrival to ICU. Not all subjects had this lab available, thus the inconsistency of numbers from the participant flow module.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sufentanil Bolus | Sufentanil Infusion
Number analyzed (Participants) | 22 | 20
ng/mL | 2.8 (0.5) | 2.8 (0.5)

ADVERSE EVENTS:
Time Frame: Procedure end time to discharge from hospital, an average of 4 days.
Description: AEs and SAEs will be captured on a source document page. AEs and SAEs will be reported to the PI within 24 hrs of notice of occurrence. AEs and SAEs will be reviewed by PI for severity and relationship.
  Any reportable AEs will be reported to the IRB within 5 business days, and SAEs will be reported to Institutional Review Board within 24 hrs of PI becoming aware of occurrence. PI will determined what follow up is needed for each event.
Arm/Group | Sufentanil Bolus | Sufentanil Infusion
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/33
Other Adverse Events (participants affected / at risk) | 4/31 | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil Bolus (N=31) | Sufentanil Infusion (N=33)
Acute left MCA stroke (Vascular disorders) | 1 (1) | 0 (0)
Emergent OR procedure (Cardiac disorders) | 0 (0) | 1 (1) — Return to OR for bleeding.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil Bolus (N=31) | Sufentanil Infusion (N=33)
Hypotension (Cardiac disorders) | 4 (4) | 5 (5) — Hypotension requiring vasopressor support in ICU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT04226495/Prot_003.pdf
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT04226495/ICF_001.pdf